CLINICAL TRIAL: NCT01982149
Title: Incorporation of Genetic Expression of Airway Epithelium With CT Screening for Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1305013973; Weill Cornell Medical College (Other Grant/Funding Number: Weill Cornell Medical College)
Record Dates: First submitted 2013-10-25; First posted 2013-11-13 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Smokers; Nonsmokers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and cells obtained for this study may be retained for future research with given consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Non-smokers (n=20)
  Interventions: Genetic: Group 1
- Group 2: Non-smokers (n=20), Smokers (n=20) and Individuals with lung cancer (n=20)
  Interventions: Genetic: Group 2
- Group 3: Subjects with abnormalities (nodules) detected on CT (n=20)
  Interventions: Genetic: Group 3

INTERVENTIONS:
Genetic: Group 1 — Perform gene expression studies of airway epithelium to correlate findings in the gene expression of nasal bronchial epithelium
  Groups: Group 1
Genetic: Group 2 — Correlate gene expression data from nasal and bronchial epithelium
  Groups: Group 2
Genetic: Group 3 — Correlated nasal epithelial gene expression with the ultimate diagnosis (by biopsy or surgery)
  Groups: Group 3

SUMMARY:
Lung cancer, largely the result of cigarette smoking, is the leading cause of cancer death in the United States, killing over 160,000 people in 2010, more than breast, colorectal, and prostate cancer combined. Since only 10% of heavy smokers develop lung cancer and 20% of lung cancers develop in nonsmokers, it is thought that genetic predisposition plays an important role. This study proposes to examine the genetic correlation between nasal and bronchial epithelium and to identify a patient's risk for lung cancer earlier.

DETAILED DESCRIPTION:
Lung cancer, largely the result of cigarette smoking, is the leading cause of cancer death in the United States, killing over 160,000 people in 2010, more than breast, colorectal, and prostate cancer combined. Since only 10% of heavy smokers develop lung cancer and 20% of lung cancers develop in nonsmokers, it is thought that genetic predisposition plays an important role.

Without screening, lung cancer is only detected at an early stage 10% of the time, translating into a 7% cure rate. Published studies of screening for lung cancer using CT scans show that it is detectable at an early stage 85% of the time, translating into a cure rate over 60%. However, in a sample population of 1000 smokers over the age of 60 (high risk individuals), 233 will have suspicious abnormalities on CT scans, but only 27 had lung cancer. Two concerns are apparent. First, among the 233 individuals with suspicious abnormalities on CT, how does one choose the ones suspicious enough for biopsy, surgery, or other invasive procedures? Generally, follow-up CT scans over several months are used to assess the abnormalities for growth, since growth is a characteristic of malignancy. Unfortunately, repeated CT scans involve financial cost and potential radiation risk. An additional technique which is able to predict predisposition to lung cancer, if combined with the ability of CT scans to detect abnormalities in real time, could prove to be a powerful platform to efficiently screen for lung cancer and reduce its mortality.

Lung cancer develops as a consequence of a series of genetic injuries to the cells lining the airways which cause these bronchial cells to grow in a malignant manner, unchecked, resistant to normal homeostatic controls. By studying the gene expression signature of airway (bronchial) lining cells, differences are observed between normal nonsmokers, individuals exposed to smoke second-hand, and smokers who have developed COPD (chronic bronchitis and emphysema). Some genetic changes in bronchial lining cells near a lung cancer are specific to lung cancer --- the "field effect." Obtaining bronchial lining cells for genetic analysis requires an invasive and expensive procedure, fiberoptic bronchoscopy, and therefore bronchoscopically acquired bronchial lining cells are not suitable for screening of the public for lung cancer.

The lining cells of the nose, the nasal epithelium, which is part of the human airway, have many similarities to bronchial epithelium, but they are much more accessible. A gentle scraping of the nasal lining involves no risk to the patient, less cost, and, it is hoped, will provide the same genetic information as the bronchial lining cells.

This study proposes to examine the genetic correlation between nasal and bronchial epithelium in the hopes of developing an office-based test to identify a patient's risk for lung cancer. It is hoped that the genetic analysis of nasal epithelium may be combined with the other risk factors for lung cancer such as cigarette smoking, age over 50 years, and an obstructive ventilatory impairment noted on pulmonary function tests to find the ideal (or enriched) population to screen with CT to detect early lung cancer, thus reducing the financial cost, radiation exposure, and risk of invasive procedures to a minimum, furthering the ultimate goal of "personalized medicine."

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* All study subjects should be able to provide informed consent
* Males or females ages 18 years and older
* Must provide HIV informed consent

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Must provide informed consent
* Males and females age 18 years and older
* Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and/or (6) diseases of organs with known association with lung disease
* Must provide HIV informed consent

Exclusion Criteria:

HEALTHY VOLUNTEER RESEARCH SUBJECTS

* Individuals not deemed in good overall health by the investigator will not be accepted into the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: - Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria).
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.
* Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.
* Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study.
* Females who are pregnant or nursing will not be accepted into the study

VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study.
* Habitual use of drugs and/or alcohol within the past six months (Acceptable: Marijuana one time in three months; average of two alcoholic beverages per day; drug and/or alcohol abuse is defined as per the DSM-IV Substance Abuse Criteria)
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Measure the correlation among gene expression levels between nasal and bronchial epithelium on an individual gene and multivariate basis | One year
  Measure the correlation among gene expression levels between nasal and bronchial epithelium on an individual gene and multivariate basis

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided